CLINICAL TRIAL: NCT05887492
Title: A Phase 1/2, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of TNG260 as Single Agent and in Combination With an Anti-PD-1 Antibody In Patients With STK11 Mutated Advanced Solid Tumors
Brief Title: Study of TNG260 and an Anti-PD Antibody in STK11 Mutated Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tango Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TNG260-C101
Record Dates: First submitted 2023-04-18; First posted 2023-06-02 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-07

CONDITIONS: Non Small Cell Lung Cancer; Solid Tumors, Adult; Lung Cancer; Lung Adenocarcinoma
Keywords: STK11; KRAS wild type; LKB1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Adenocarcinoma of Lung | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Phase 1 (Dose Escalation) and Phase 2 (Dose Expansion)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation (Experimental): Participants with STK11-mutant solid tumors will receive escalating doses of TNG260 in combination with pembrolizumab to estimate the MTD
  Interventions: Drug: TNG260; Drug: Pembrolizumab
- Dose Expansion in NSCLC with KRAS Mutation (Experimental): Participants with STK11-mutant and KRAS-mutant NSCLC (squamous and non squamous) will receive TNG260 at the identified RP2D in combination with pembrolizumab
  Interventions: Drug: TNG260; Drug: Pembrolizumab
- Dose Expansion in NSCLC with KRAS Wild type (Experimental): Participants with STK11-mutant and KRAS-wild type NSCLC (squamous and non-squamous) will receive TNG260 at the identified RP2D in combination with pembrolizumab
  Interventions: Drug: TNG260; Drug: Pembrolizumab
- Dose Expansion in Advanced or Metastatic Solid Tumors (Experimental): Participants with STK11-mutant solid tumors (including but not limited to pancreatic, endometrial, cervical, breast, and carcinoma of unknown primary) will receive TNG260 at the identified RP2D in combination with pembrolizumab
  Interventions: Drug: TNG260; Drug: Pembrolizumab

INTERVENTIONS:
Drug: TNG260 — CoREST inhibitor, administered orally
Drug: Pembrolizumab — Pembrolizumab, an anti-PD-1 antibody, administered intravenously
  Other Names: Keytruda

SUMMARY:
The goal of this interventional clinical trial is to learn about TNG260, a CoREST inhibitor, in combination with pembrolizumab in patients with advanced solid tumors with a known STK11 mutation.

The main question[s] it aims to answer are:

* the recommended dose for Phase 2
* to evaluate the safety and tolerability of the combination therapy
* to determine the pharmacokinetics of TNG260
* to evaluate the initial antineoplastic activity

Participants will receive study treatment until they experience an undesirable side effect, their disease progresses or until they withdraw consent.

DETAILED DESCRIPTION:
This is a first-in-human Phase 1/2, open-label, multicenter, dose-escalation and expansion study designed to determine the maximum tolerated dose and recommended phase 2 dose(s) and evaluate the safety and tolerability, pharmacokinetics, and antineoplastic activity of escalating oral doses of TNG260 when administered with a standard dose of pembrolizumab in participants with locally advanced or metastatic STK11 mutated solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Is ≥18 years of age at the time of signature of the main study ICF.
* Has ECOG performance status of 0 or 1.
* Has measurable disease based on RECIST v1.1.
* All participants must have documented STK11 mutation in a solid tumor, which is identified through a validated analytical method
* Has confirmed histologic or cytologic diagnosis of a locally advanced or metastatic solid tumor.
* Adequate organ function/reserve per local labs
* Adequate liver function per local labs
* Adequate renal function per local labs
* Negative serum pregnancy test result at screening
* Written informed consent must be obtained according to local guidelines

Exclusion Criteria:

* Known allergies, hypersensitivity, or intolerance to TNG260, PD-1 antibody or its excipients
* Uncontrolled intercurrent illness that will limit compliance with the study requirements
* Active infection requiring systemic therapy
* Currently participating in or has planned participation in a study of another investigational agent or device
* Impairment of GI function or disease that may significantly alter the absorption of oral TNG260
* Active prior or concurrent malignancy.
* Central nervous system metastases associated with progressive neurological symptoms
* Current active liver disease from any cause
* Clinically relevant cardiovascular disease
* A female patient who is pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Determine the MTD and RP2D(s) (Phase 1 only) | 42 days
  To determine the MTD and RP2D(s) of TNG260 when administered in combination with pembrolizumab
Measure antitumor activity using RECIST 1.1 (Phase 2 only) | 12 weeks
  To assess antineoplastic activity of TNG260 when administered in combination with pembrolizumab in participants with locally advanced unresectable or metastatic STK11-mutated solid tumors by measuring ORR, DOR, and PFS by RECIST 1.1

SECONDARY OUTCOMES:
Measure antitumor evidence of TNG260 + pembrolizumab antineoplastic activity by RECIST 1.1 (Phase 1 only) | 12 weeks
  To assess antineoplastic activity of TNG260 when administered in combination with pembrolizumab in participants with locally advanced unresectable or metastatic STK11-mutated solid tumors by measuring ORR, DOR, and PFS by RECIST 1.1
Characterize Area Under the Curve (AUC) of TNG260 | 37 days
  Measure the plasma concentration versus time curve (AUC) of TNG260 alone and when administered in combination with pembrolizumab
Characterize the time to achieve Time to Maximal Concentration (Tmax) of TNG260 | 37 days
  To characterize the Tmax by measuring the plasma concentrations versus time of TNG260 alone and when administered in combination with pembrolizumab
Characterize Maximum Observed Plasma Concentration (Cmax) of TNG260 | 37 days
  To characterize the Cmax by measuring the plasma concentrations versus time of TNG260 alone and when administered in combination with pembrolizumab
Characterize Terminal Half-life (T1/2) of TNG260 | 37 days
  To characterize the T1/2 by measuring the plasma concentrations versus time of TNG260 alone and when administered in combination with pembrolizumab
Characterize pembrolizumab concentrations when administered with TNG260 | 43 days
  To characterize the pre treatment and trough concentration levels of pembrolizumab when administered in combination with TNG260
Safety and tolerability of TNG260 by CTCAE 5.0 | 42 days
  To evaluate the safety and tolerability of TNG260 when administered as single agent and in combination with pembrolizumab by measuring the incidence, nature, and severity of AE and SAE graded according to CTCAE v5.0
To measure changes in histone acetylation when administered with TNG260 | 12 weeks
  Measure changes in levels of histone acetylation in blood and/or tumor tissue, on study treatment relative to pre-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Adam Crystal, MD, PhD, Study Director — Tango Therapeutics, Inc.
Locations (13):
- United States (13):
  - UCLA Hematology/Oncology, Santa Monica, California
  - SCRI at HealthOne, Denver, Colorado
  - Florida Cancer Specialists, Sarasota, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - START MidWest, Grand Rapids, Michigan
  - NYU Langone Hematology Oncology Associates-Mineola, Mineola, New York
  - New York University Langone Health, New York, New York
  - Sarah Cannon Tennessee Oncology, Nashville, Tennessee
  - US Oncology Investigational Products Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology Virginia, Fairfax, Virginia
  - US Oncology Investigational Products Center, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No